CLINICAL TRIAL: NCT00334282
Title: A Randomised, Double-blind, Placebo Controlled, Multi-center Phase III Study to Evaluate the Efficacy and Safety of Pazopanib (GW786034) Compared to Placebo in Patients With Locally Advanced and/or Metastatic Renal Cell Carcinoma
Brief Title: Safety and Efficacy of GW786034 (Pazopanib) In Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VEG105192
Record Dates: First submitted 2006-06-05; First posted 2006-06-07 (Estimated); Results first posted 2010-08-02 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2015-08

CONDITIONS: Carcinoma, Renal Cell
Keywords: Metastatic; Anti-angiogenesis; GW786034; Pazopanib
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo arm (Placebo Comparator): matching placebo (800 mg tablet) once daily
  Interventions: Drug: placebo
- pazopanib arm (Experimental): Oral pazopanib tablet 800 mg once daily continuously
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Oral pazopanib tablet 800 mg once daily continuously
  Other Names: votrient
  Arms: pazopanib arm
Drug: placebo — matching placebo (800 mg tablet) once daily
  Arms: placebo arm

SUMMARY:
To evaluate efficacy and safety of pazopanib compared to placebo in patients with locally advanced and/ or metastatic renal cell carcinoma (RCC). Approximately 350-400 eligible patients will be stratified and randomized in a 2:1 ratio to receive either 800 mg pazopanib once daily or matching placebo. The study treatment will continue until patients experience disease progression, unacceptable toxicity or death. Primary objective of the study is to evaluate and compare the two treatment arms for progression-free survival. Principal secondary objective is to evaluate and compare the two treatment arms with respect to overall survival. Other objectives are overall response rate [complete response (CR) + partial response (PR)], rate of CR + PR + 6 months stable disease, and the incidence, severity and causality of adverse events and serious adverse events. Safety and efficacy assessments will be regularly performed on all patients. An Independent Data Monitoring Committee will be established to monitor safety during the course of the study and to evaluate interim efficacy data on overall survival.

ELIGIBILITY:
Inclusion Criteria:

A patient will be considered for inclusion in this study only if all of the following criteria apply:

* Signed written informed consent.
* Diagnosis of clear cell RCC that is predominantly clear cell histology. Note: cytology cannot be the only pathologic criteria to confirm clear cell RCC. Patients with tumor types that are interpreted as non-clear cell, e.g. papillary, are excluded.
* Locally advanced RCC (defined as disease not amenable to curative surgery or radiation therapy) or metastatic RCC (equivalent to Stage IV RCC according to American Joint Committee on Cancer (AJCC) staging.
* Note: If the metastatic disease is restricted to a solitary lesion, its neoplastic nature must be confirmed by histology or cytology. Cytology cannot be the only pathologic criteria to confirm clear cell RCC, but can be used in a patient with histologically confirmed clear cell RCC to confirm that metastatic disease is neoplastic in nature.
* Must have measurable disease, i.e. presenting with at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST). A measurable lesion is defined as a lesion that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques, or ≥ 10 mm with spiral CT scan.
* Note: Patient should be excluded if all baseline measurable lesions are within previously irradiated areas.
* Note: A patient must complete all the baseline disease assessments in order to be eligible. Baseline head, chest, abdominal and pelvic CT or MRI scans must be performed within 2 weeks prior to the first dose of study medication; baseline bone scan must be performed within 3 weeks of the first dose of study medication.
* Patients who have received only one prior systemic treatment for locally advanced or metastatic RCC with documented disease progression or documented treatment discontinuation due to unacceptable toxicity. This first-line systemic treatment must be cytokine based.
* Note: The first-line cytokine-based treatment can be interleukin-2 (IL-2) or interferon-α (INFα) monotherapy, IL-2 in combination with INF-α, IL-2 and/or INF-α in combination with chemotherapy, hormonal or other therapies excluding agents targeting angiogenesis pathways. Agents in a combination regimen can be given sequentially if the treatment sequence is pre-determined and the patient does not fail one agent prior to starting another.
* Note: Prior adjuvant or neo-adjuvant therapies are permitted excluding any agents that target vascular endothelial growth factor (VEGF) or VEGF receptors. The adjuvant/neo-adjuvant therapies should not be considered as first-line systemic treatment for advanced RCC.

Or,

* Patients who have received no prior systemic therapy for advanced/metastatic RCC can be enrolled if under any of the following circumstances:
* Patients who live in countries or regions where there is no established standard first-line therapy for advanced/metastatic RCC or where there are barriers to the access of established therapies such as sunitinib, sorafenib, IFNα or IL-2.
* Patients who live in countries or regions where IL-2 or INF-α has been approved for the treatment of advanced/metastatic RCC, however, these agents are generally not recognized by the local clinical community as a standard treatment for advanced/metastatic RCC, or where the physician and the patient have determined that the available cytokine therapies are not an acceptable therapeutic option.
* Patients who have recurred following prior adjuvant or neo-adjuvant cytokine therapy for RCC are eligible to participate without receiving a first-line systemic treatment for locally advanced or metastatic RCC. These patients should be stratified as the first-line population.
* Male or female ≥ 18 years of age.
* A woman is eligible to participate in the study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:
* Has had a hysterectomy,
* Has had a bilateral oophorectomy (ovariectomy),
* Has had a bilateral tubal ligation,
* Is post-menopausal (total cessation of menses for ≥1 year).
* Childbearing potential, has a negative serum pregnancy test within 2 weeks of the first dose of study medication, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:
* An intrauterine device with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the female patient's entry and is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigation product, through the clinical trial, and for at least 21 days after the last dose of investigational product.
* Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).
* Oral contraceptives are not reliable due to the potential for drug-drug interactions.
* A man with a female partner of childbearing potential is eligible to enter and participate in the study if he is abstinent or uses a barrier method of contraception during the study.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1
* Adequate baseline organ function defined as:
* Hematologic function:

Absolute Neutrophil Count (ANC) ≥1 x 10^9/L Hemoglobin ≥ 9 g/dL Platelet ≥75 x 10^9/L

* Hepatic function:

Total bilirubin ≥ 1.5 x Upper Limit of Normal (ULN) Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≥ 2 x ULN

* Renal function:

Calculated creatinine clearance≥30 mL/min [See Section 14.6 Appendix 6] and

≥Urine protein is 0, trace, or +1 determined by dipstick urinalysis, or < 1.0 gram determined by 24-hour urine protein analysis.

* Note: A patient should first be screened with dipstick urinalysis. If urine protein is ≥2+, then a 24-hour urine protein must be assessed and patient will be excluded if 24-hour urine protein is≥ 1.0 gram.
* Corrected serum calcium level within normal range per local clinical laboratory standard.

Note: Patients with hypercalcemia should be treated until the corrected serum calcium level reaches the normal range.

* At least 4 weeks must have elapsed since the last surgery and 2 weeks must have elapsed since radiotherapy or the last systemic cytokine therapy.
* Complete recovery from prior surgery, and/or reduction of all AEs to Grade 1 from prior systemic therapy or radiotherapy.
* Note: In patients with prior radiotherapy, the steroid doses should be stable or decreasing for at least 2 weeks.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

* Pregnant or lactating female.
* History of another malignancy.
* Note: Patients who have had another malignancy and have been disease-free for 5 years, or patients with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* History or presence of central nervous system (CNS) metastasis or leptomeningeal tumors as documented by CT or MRI scan, analysis of cerebrospinal fluid or neurological exam.

Note: A baseline brain CT or MRI scan must be obtained in all patients within 2 weeks of the first dose of study medication.

* Malabsorption syndrome or disease that significantly affects gastrointestinal function, or major resection of the stomach or small bowel that could affect the absorption of pazopanib.
* Unable to swallow and retain orally administered medication.
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to beginning study treatment.
* History of human immunodeficiency virus infection.
* Presence of uncontrolled infection.
* Corrected QT interval (QTc) prolongation defined as QTc interval > 470 msecs.
* History of Class III or IV congestive heart failure according to New York Heart Association (NYHA) classification.
* History of any one of the following cardiac conditions within the past 6 months:
* Cardiac angioplasty or stenting, or
* Myocardial infarction, or
* Unstable angina.
* History of cerebrovascular accident within the past 6 months.
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140mmHg, or diastolic blood pressure (DBP) of ≥ 90mmHg].
* Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. The blood pressure must be re-assessed on two occasions that are separated by a minimum of 24 hours. The mean SBP / DBP values from both blood pressure assessments must be < 140/90mmHg in order for a patient to be eligible for the study.
* History of untreated deep venous thrombosis (DVT) within the past 6 months (e.g. a calf vein thrombosis that is not treated).

Note: Patients with recent DVT who are treated with therapeutic anti-coagulating agents (excluding therapeutic warfarin) for at least 2 weeks are eligible.

* Presence of any non-healing wound, fracture, or ulcer, or presence of symptomatic peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with patient's safety, obtaining informed consent or compliance to the study.
* Has taken any prohibited medications within 14 days of the first dose of study medication.
* Current or prior use of an investigational anti-cancer drug within 4 weeks of start of study.
* Prior use of an investigational or licensed drug that targets VEGF or VEGF receptors (eg. bevacizumab, sunitinib, sorafenib, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2006-04; Primary Completion 2008-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (85):
- Argentina (5):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (5):
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Wodonga, Victoria
- Austria (2):
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Brazil (3):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Jaú, São Paulo
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, Beijing, China
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Chomutov
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Prague
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Thessaloniki
- Hong Kong (3):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Tuen Mun, New Territories
- India (5):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Trivandrum
- Ireland (2):
  - GSK Investigational Site, Galway
  - GSK Investigational Site, Tallaght, Dublin
- Italy (6):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Casalpusterlengo (LO), Lombardy
  - GSK Investigational Site, Crema, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Orbassano (TO), Piedmont
- GSK Investigational Site, Riga, Latvia
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Mexico City
- New Zealand (3):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Newtown, Wellington
  - GSK Investigational Site, Palmerston North
- Pakistan (3):
  - GSK Investigational Site, Islamabad
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- Poland (5):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Russia (8):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- GSK Investigational Site, Bratislava, Slovakia
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Songpa-gu, Seoul
- Tunisia (3):
  - GSK Investigational Site, Sfax
  - GSK Investigational Site, Sousse
  - GSK Investigational Site, Tunis
- Ukraine (5):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Zaporizhzhya
- United Kingdom (5):
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Bebington, Wirral
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Swansea

REFERENCES:
- [Background] Bonate PL, Suttle AB. Modeling tumor growth kinetics after treatment with pazopanib or placebo in patients with renal cell carcinoma. Cancer Chemother Pharmacol. 2013 Jul;72(1):231-40. doi: 10.1007/s00280-013-2191-0. Epub 2013 May 29. PMID 23715625
- [Background] Tran HT, Liu Y, Zurita AJ, Lin Y, Baker-Neblett KL, Martin AM, Figlin RA, Hutson TE, Sternberg CN, Amado RG, Pandite LN, Heymach JV. Prognostic or predictive plasma cytokines and angiogenic factors for patients treated with pazopanib for metastatic renal-cell cancer: a retrospective analysis of phase 2 and phase 3 trials. Lancet Oncol. 2012 Aug;13(8):827-37. doi: 10.1016/S1470-2045(12)70241-3. Epub 2012 Jul 2. PMID 22759480
- [Background] Sternberg CN, Davis ID, Mardiak J, Szczylik C, Lee E, Wagstaff J, Barrios CH, Salman P, Gladkov OA, Kavina A, Zarba JJ, Chen M, McCann L, Pandite L, Roychowdhury DF, Hawkins RE. Pazopanib in locally advanced or metastatic renal cell carcinoma: results of a randomized phase III trial. J Clin Oncol. 2010 Feb 20;28(6):1061-8. doi: 10.1200/JCO.2009.23.9764. Epub 2010 Jan 25. PMID 20100962
- [Background] Maitland ML, Wu K, Sharma MR, Jin Y, Kang SP, Stadler WM, Karrison TG, Ratain MJ, Bies RR. Estimation of renal cell carcinoma treatment effects from disease progression modeling. Clin Pharmacol Ther. 2013 Apr;93(4):345-51. doi: 10.1038/clpt.2012.263. Epub 2012 Dec 27. PMID 23443753
- [Background] Xu CF, Reck BH, Goodman VL, Xue Z, Huang L, Barnes MR, Koshy B, Spraggs CF, Mooser VE, Cardon LR, Pandite LN. Association of the hemochromatosis gene with pazopanib-induced transaminase elevation in renal cell carcinoma. J Hepatol. 2011 Jun;54(6):1237-43. doi: 10.1016/j.jhep.2010.09.028. Epub 2011 Feb 12. PMID 21145803
- [Background] Xu CF, Reck BH, Xue Z, Huang L, Baker KL, Chen M, Chen EP, Ellens HE, Mooser VE, Cardon LR, Spraggs CF, Pandite L. Pazopanib-induced hyperbilirubinemia is associated with Gilbert's syndrome UGT1A1 polymorphism. Br J Cancer. 2010 Apr 27;102(9):1371-7. doi: 10.1038/sj.bjc.6605653. Epub 2010 Apr 13. PMID 20389299
- [Background] Sternberg CN, Hawkins RE, Wagstaff J, Salman P, Mardiak J, Barrios CH, Zarba JJ, Gladkov OA, Lee E, Szczylik C, McCann L, Rubin SD, Chen M, Davis ID. A randomised, double-blind phase III study of pazopanib in patients with advanced and/or metastatic renal cell carcinoma: final overall survival results and safety update. Eur J Cancer. 2013 Apr;49(6):1287-96. doi: 10.1016/j.ejca.2012.12.010. Epub 2013 Jan 12. PMID 23321547
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Goldstein D, Rosenberg JE, Figlin RA, Townsend RR, McCann L, Carpenter C, Pandite L. Is change in blood pressure a biomarker of pazopanib and sunitinib efficacy in advanced/metastatic renal cell carcinoma? Eur J Cancer. 2016 Jan;53:96-104. doi: 10.1016/j.ejca.2015.10.006. Epub 2015 Dec 15. PMID 26702763
- [Derived] Sorich MJ, Kichenadasse G, Rowland A, Woodman RJ, Mangoni AA. Angiotensin system inhibitors and survival in patients with metastatic renal cell carcinoma treated with VEGF-targeted therapy: A pooled secondary analysis of clinical trials. Int J Cancer. 2016 May 1;138(9):2293-9. doi: 10.1002/ijc.29972. Epub 2016 Jan 6. PMID 26685869
- [Derived] Suttle AB, Ball HA, Molimard M, Hutson TE, Carpenter C, Rajagopalan D, Lin Y, Swann S, Amado R, Pandite L. Relationships between pazopanib exposure and clinical safety and efficacy in patients with advanced renal cell carcinoma. Br J Cancer. 2014 Nov 11;111(10):1909-16. doi: 10.1038/bjc.2014.503. Epub 2014 Oct 28. PMID 25349968

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib 800 mg: Pazopanib 800 mg (tablets) administered orally once a day
- Placebo: Matching Placebo administered orally once a day
Period: Overall Study
Arm/Group | Pazopanib 800 mg | Placebo
Started | 290 | 145
Completed | 68 | 37
Not Completed | 222 | 108
Not completed — Lost to Follow-up | 11 | 5
Not completed — Withdrawal by Subject | 17 | 3
Not completed — Death | 194 | 100

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matching Placebo administered once a day
- Total: Total of all reporting groups
Arm/Group | Pazopanib 800 mg | Placebo | Total
Number analyzed (Participants) | 290 | 145 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.06) | 59.6 (11.04) | 59.3 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 36 | 128
  Male | 198 | 109 | 307
Race/Ethnicity, Customized [Number; unit: participants]
  White | 252 | 122 | 374
  Asian | 36 | 23 | 59
  African American/African Heritage | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the interval between the date of randomization and the earliest date of disease progression or death due to any cause. Assessments of progression and non-progression were made by an independent imaging review committee (IRC) for the primary analysis.
Time Frame: Randomization until progression (up to 2 years)
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib 800 mg | Placebo
Number analyzed (Participants) | 290 | 145
months | 9.2 [7.4 to 12.9] | 4.2 [2.8 to 5.6]
Statistical Analysis 1: Comparison: Pazopanib 800 mg; Test type: Superiority or Other; p = .0000001, Log Rank — stratified log-rank test; Hazard Ratio (HR) = 0.46, 95% CI [0.34 to 0.62] — The estimated value is the hazard ratio comparing pazopanib to placebo

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death. The length of this interval was estimated as the date of death minus the date of randomization plus 1 day. Participants who were still alive at the time of analysis were censored.
Time Frame: Randomization until death (up to 2 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib 800 mg | Placebo
Number analyzed (Participants) | 290 | 145
months | 22.9 [19.9 to 25.4] | 20.5 [15.6 to 27.6]

3. Secondary Outcome: Overall Response
Description: Overall response is the number of participants who had a complete response (CR) or a partial response (PR). Per RECIST: CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the Baseline sum, no worsening of non-TLs, and no new lesions; Progressive disease (PD), a >=20% increase in TLs, clearly worsening of non-TLs, or emergence of new lesions; Stable Disease, small changes that do not meet previously given criteria. IRC, independent review committee.
Time Frame: Baseline until either response or progression (up to 2 years)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg | Placebo
Number analyzed (Participants) | 290 | 145
participants
  Complete Response, IRC assessed | 1 | 0
  Partial Response, IRC assessed | 87 | 5
  Stable Disease, IRC assessed | 110 | 59
  Progressive Disease, IRC assessed | 51 | 58
  Unknown, IRC assessed | 41 | 23
  Complete Response, Investigator assessed | 4 | 0
  Partial Response, Investigator assessed | 99 | 9
  Stable Disease, Investigator assessed | 118 | 62
  Progressive Disease, Investigator assessed | 46 | 65
  Unknown, Investigator assessed | 23 | 9

4. Secondary Outcome: Participants With Complete Response, Partial Response, or 6 Months of Stable Disease
Description: This is similar to overall response rate, but also includes participants who had stable disease for at least 6 months. Per Response Evaluation Criteria In Solid Tumors (RECIST): CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the Baseline sum; Stable Disease, small changes that do not meet previously given criteria; Progressive Disease, a >=20% increase in target lesions. IRC, independent review committee.
Time Frame: Baseline until 6 months post-Baseline or progressive disease
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg | Placebo
Number analyzed (Participants) | 290 | 145
participants
  Complete Response, IRC assessed | 1 | 0
  Partial Response, IRC assessed | 87 | 5
  6 Months Stable Disease, IRC assessed | 48 | 17
  Progressive Disease, IRC assessed | 92 | 84
  Unknown | 62 | 39

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from first observation of response until progression of disease or death.
Time Frame: Time from response until progression (up to 2 years)
Population: ITT Population. Only results for pazopanib are given because there were not enough placebo responders.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 290
weeks | 58.7 [52.1 to 68.1]

6. Secondary Outcome: Time to Response as Assessed by an Independent Review Committee (IRC) and the Investigator
Description: Time to response is defined as the time from randomization until the first documented evidence of complete response (all detectable tumor has disappeared) or partial response (a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the Baseline sum) (whichever status was recorded first).
Time Frame: Randomization until CR or PR (assessed for up to 2 years)
Population: ITT Population. Only participants with a complete or partial response were analyzed. Only results for pazopanib are given because there were not enough placebo responders. The different number of participants analyzed is due to differences in clinical judgement, measurement, and the selection of target lesions.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 103
weeks
  IRC assessed, n=88 | 11.9 [9.4 to 12.3]
  Investigator assessed, n=103 | 12.0 [11.6 to 12.3]

7. Secondary Outcome: Adjusted Mean Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life (QOL) Questionnaire Core 30 (EORTC QLQ C-30) Score at Weeks 6, 12, 18, 24, and 48
Description: The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer participants. The analyses for EORTC QLQ-C30 were focused on global health status/Health-Related Quality of Life (HRQOL) scores on the questionnaire. The scores (from 1 [very poor quality of life] to 7 [excellent quality of life]) for these two questions were averaged and then transformed to a 0 - 100 scale (based on published methods) prior to analysis of change from Baseline.
Time Frame: Baseline and Weeks 6, 12, 18, 24, and 48
Population: Participants in the ITT Population who completed HRQOL assessments at Baseline and had at least one post-Baseline assessment are included. Only participants who were on treatment at the given time point were asked to complete the questionnaire, and only those who completed the questionnaire could be analyzed for each individual time point.
Measure: Mean (Standard Deviation); unit: points on a scale
Groups:
- Pazopanib: Pazopanib 800 mg (tablets) administered orally once a day
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 246 | 111
points on a scale
  Week 6, n=243, 110 | -3.2 (19.66) | -2.6 (19.18)
  Week 12, n=219, 81 | -3.6 (20.16) | -0.5 (17.55)
  Week 18, n=191, 61 | -2.5 (21.70) | -0.3 (18.13)
  Week 24, n=164, 49 | 0.1 (19.81) | -0.5 (18.67)
  Week 48, n=96, 24 | -0.3 (18.36) | 0.3 (15.63)

8. Secondary Outcome: Adjusted Mean Change From Baseline in the Index Score of the EQ-5D (EuroQoL [Quality of Life]-5D) Questionnaire at Weeks 6, 12, 18, 24, and 48
Description: The EQ-5D is comprised of a 5-item health status measure and a visual analogue rating scale, and measures mobility, self-care, usual activities, pain, discomfort, and anxiety/depression. Responses to each of the 5 health states are measured on a 3-point scale (no, moderate, and extreme problems). Scoring of the EQ-5D yields an index-based summary score (Index), through application of societal weights, and a VAS score (VAS). Index is interpreted on a continuum from 1.0 (best possible health) to 0 (represents dead), to some health sates being worse than dead (<0).
Time Frame: Baseline and Weeks 6, 12, 18, 24, and 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Pazopanib 800 mg | Placebo
Number analyzed (Participants) | 253 | 125
points on a scale
  Week 6, n=253, 125 | -0.014 (0.2203) | -0.029 (0.2674)
  Week 12, n=219, 86 | -0.040 (0.2148) | 0.007 (0.1969)
  Week 18, n=196, 62 | -0.023 (0.2305) | -0.006 (0.1466)
  Week 24, n=166, 51 | -0.025 (0.2420) | -0.001 (0.2411)
  Week 36, n=98, 24 | 0.030 (0.1961) | -0.005 (0.2015)

9. Secondary Outcome: Adjusted Mean Change From Baseline in the Visual Analog Scale (VAS) Score of the EQ-5D (EuroQoL [Quality of Life]-5D) Questionnaire at Weeks 6, 12, 18, 24, and 48
Description: The EQ-5D is comprised of a 5-item health status measure and a visual analogue rating scale, and measures mobility, self-care, usual activities, pain, discomfort, and anxiety/depression. Responses to each of the 5 health states are measured on a 3-point scale (no, moderate, and extreme problems). Scoring of the EQ-5D yields an index-based summary score (Index) and a VAS score (VAS), obtained from participant's self-reports of their health on a VAS thermometer scale. The EQ-5D VAS ranges from 0% (worst imaginable health state) to 100% (best imaginable health state).
Time Frame: Baseline and Weeks 6, 12, 18, 24, and 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Pazopanib 800 mg | Placebo
Number analyzed (Participants) | 239 | 111
points on a scale
  Week 12, n=212, 80 | -0.9 (21.07) | -3.6 (23.04)
  Week 6, n=239, 111 | 0.4 (22.55) | 0.2 (25.35)
  Week 18, n=189, 60 | 0.1 (23.20) | 0.1 (19.35)
  Week 24, n=161, 49 | 2.6 (22.16) | 5.4 (21.27)
  Week 36, n=95, 23 | 2.4 (24.21) | 8.8 (23.96)

10. Secondary Outcome: Plasma Pazopanib Concentrations Before Dosing and at 2, 4, and 8 Hours After Dosing on Day 1 and Week 3
Description: The concentration of pazopanib in the plasma was measured.
Time Frame: Day 1 and Week 3
Population: Subgroup of enrolled participants who agreed to have blood samples collected for analysis of pazopanib in plasma. Data were missing or not collected at Week 3 for 8 participants for whom data were available on Day 1. No samples were collected at Week 3 from 2 participants.
Measure: Median (Full Range); unit: nanograms per milliliter
Groups:
- Pazopanib 800 mg: Pazopanib 800 mg (tablets) administered once daily
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 57
nanograms per milliliter
  Day 1, before dosing, n=57 | 0 [0 to 846]
  Week 3, before dosing, n=48 | 31851 [2634 to 61720]
  Day 1, 2 hours after dosing, n=57 | 17270 [0 to 107454]
  Week 3, 2 hours after dosing, n=49 | 42205 [4282 to 79977]
  Day 1, 4 hours after dosing, n=57 | 24360 [2371 to 74606]
  Week 3, 4 hours after dosing, n=49 | 42637 [3532 to 107972]
  Day 1, 8 hours after dosing, n=57 | 19925 [3273 to 60974]
  Week 3, 8 hours after dosing, n=48 | 40177.5 [3760 to 96548]

11. Secondary Outcome: Baseline Expression Levels of the Indicated Target Proteins in Pazopanib- and Placebo-treated Participants
Description: Baseline plasma samples were obtained from participants and were tested for the indicated cytokine and angiogenesis factors. Protein levels were determined using the Searchlight multiplex system based on chemiluminescence.
Time Frame: Baseline
Population: Subgroup of enrolled participants who agreed to have plasma samples collected for biomarker analyses.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Pazopanib 800 mg | Placebo
Number analyzed (Participants) | 225 | 119
picograms per milliliter
  Interleukin-6 | 31.003 (65.247) | 24.145 (31.708)
  Interleukin-8 | 35.429 (164.12) | 27.755 (66.129)
  Vascular endothelial growth factor | 308.61 (365.19) | 273.15 (350.91)
  Hepatocyte growth factor | 383.55 (308.89) | 522.94 (1003.8)
  Tissue inhibitor of metalloproteinase 1 | 847464 (690744) | 735915 (423493)
  e-Selectin | 41649.28 (22389.04) | 41231.45 (19825.7)
  Osteopotin | 444343 (707005) | 369317 (490931)

ADVERSE EVENTS:
Time Frame: Date of study entry until 28 days after the last dose.
Arm/Group | Pazopanib 800 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 79/290 | 28/145
Other Adverse Events (participants affected / at risk) | 258/290 | 87/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=290) | Placebo (N=145)
Diarrhea (Gastrointestinal disorders) | 6 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1
Hepatotoxicity (Hepatobiliary disorders) | 3 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Paraplegia (Nervous system disorders) | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Coordination abnormal (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Myelitis (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Alanine aminotransferase increasead (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Skin graft failure (Injury, poisoning and procedural complications) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anorectal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=290) | Placebo (N=145)
Diarrhoea (Gastrointestinal disorders) | 149 | 13
Nausea (Gastrointestinal disorders) | 75 | 13
Vomiting (Gastrointestinal disorders) | 59 | 12
Abdominal pain (Gastrointestinal disorders) | 32 | 2
Abdominal pain upper (Gastrointestinal disorders) | 24 | 8
Constipation (Gastrointestinal disorders) | 20 | 9
Hair colour changes (Skin and subcutaneous tissue disorders) | 109 | 5
Rash (Skin and subcutaneous tissue disorders) | 24 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 17 | 1
Fatigue (General disorders) | 58 | 13
Asthenia (General disorders) | 44 | 13
Pyrexia (General disorders) | 14 | 9
Hypertension (Vascular disorders) | 115 | 16
Alanine aminotransferase increased (Investigations) | 54 | 4
Aspartate aminotransferase increased (Investigations) | 46 | 5
Weight decreased (Investigations) | 31 | 6
Decreased appetite (Metabolism and nutrition disorders) | 70 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 9
Headache (Nervous system disorders) | 31 | 8
Dysgeusia (Nervous system disorders) | 25 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 2
Proteinuria (Renal and urinary disorders) | 30 | 0
Insomnia (Psychiatric disorders) | 16 | 10
Hypothyroidism (Endocrine disorders) | 20 | 0
Dyspepsia (Gastrointestinal disorders) | 17 | 1
Chest pain (General disorders) | 16 | 2
Neutropenia (Blood and lymphatic system disorders) | 15 | 0
Anaemia (Blood and lymphatic system disorders) | 19 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.